CLINICAL TRIAL: NCT01229774
Title: Use of Etoricoxib Compared to Diclofenac in the Perioperative Treatment of Patients After Total Hip Arthroplasty, a Prospective, Double Blind, Phase III Study
Brief Title: Use of Etoricoxib Compared to Diclofenac in the Perioperative Treatment of Patients After Total Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Joachim Grifka, MD, Professor, Department of Orthopedic Surgery, Bad Abbach
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Eto-Dic-01
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Coxarthrosis; Arthroplasties Hip Replacement; Perioperative Blood Loss
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Etoricoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib (Experimental)
  Interventions: Drug: Etoricoxib
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Etoricoxib — Arcoxia 90 mg once a day in the evening day -1 and 0 and once a day in the morning days 1-7 plus on tablett of placebo every evening
  Arms: Etoricoxib
Drug: Diclofenac — Voltaren Resinat 75mg once a day on day -1 and 0 in the evening; twice a day (in the morning and in the evening) days 1-7
  Arms: Diclofenac

SUMMARY:
The primary aim of this study is to test if etoricoxib decreases the perioperative blood loss compared to diclofenac.

Secondary questions to be explored are:

* Does etoricoxib prevent Heterotopic ossification after Total Hip Arthroplasty as well as diclofenac ?
* Do diclofenac and etoricoxib both reduce pain at rest and on movements?
* Does etoricoxib compared to diclofenac reduce the amount of rescue medication (Oxycodon)?
* Does etoricoxib improve gastrointestinal tolerability compared to diclofenac?

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) is a common surgical procedure in orthopaedic surgery which can be associated with perioperative blood loss and severe postoperative pain. Adequate pain management is very important to achieve early mobilisation in order to avoid immobility-induced complications. Non steroidal antirheumatic agents (NSAIDs) as selective Cox-2 inhibitors are commonly used in the management of postoperative pain. There exist non-selective and selective Cox-inihibitors. Non-selective NSAIDs block the systhesis of prostagandins by the two iso-enzymes of the cyclooxygenase, Cox-1 and Cox-2. For this reason the bleeding risk after operations (e.g.tonsillectomy) is increased.

In this regard, the perioperative use of Cox-2 selective NSAIDs is advantageous for pain management after tonsillectomy. This could be shown for Rifecoxib, a selective Cox-2 inihibitor. For THAs with treatment of Etoricoxib, also a selective Cox-2 inhibitor, possible complications as the increased risk of haematoma, gastrointestinal bleeding and the need of blood transfusion could possibly be reduced. Selective Cox-2 inhibitors do not interfere with the coagulation system. Study results show that other selective Cox-2 inhibitors like meloxicam reduce perioperative blood loss. Thus, besides ensuring a good perioperative pain management, selective Cox-2 inhibitors may in addition cause less blood loss than non-selective NSAIDs.This possible reduction of blood loss during pain management with Etoricoxib (Arcoxia) will be investigated the described clinical trial.

Heterotopic ossification (HO) is a complication occurring after THA which can lead to postoperative pain and reduced function. Non-selective NSAIDs are commonly used in the prophylaxis of heterotopic ossifications after THA. The exact mechanism of prevention of bone formation is unclear. Some results indicate that the development of HO follows a Cox-2 pathway. A further aim of this clinical trial is to investigate the efficacy of Etoricoxib in the prevention of heterotropic ossification.

ELIGIBILITY:
Inclusion Criteria:

* Indication for THA because of primary and secondary osteoarthritis of the hip.
* male or female patients of the age of 55 - 85 years
* informed consent afer having been informed in detail about the clinical trial by the investigator
* negative pregnancy test (<= 2 days before inclusion) for women with child bearing potential (pre menopausal, <2 years menopausal, not surgically sterile), use of high security contraception methods as oral contraception agents or preservatives. The use of high security conception methods is also to obligatory for male patients

Exclusion Criteria:

* Known hypersensitivity to one of the two investigational medical products or substaces of similar chemical structure or to any of the excipients
* Patients who have experienced bronchospasm, asthma, acute rhinitis, urticaria, or allergic-type reactions after taking acetylsalicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors
* unexplained dysfunction of haematopoiesis
* treatment with NSAIDs or coxiben in the past 5 days before start of study
* Active peptic ulceration or active gastro-intestinal (GI) bleeding
* Pregnancy and lactation
* Congestive heart failure (NYHA II-IV)
* Established ischaemic heart disease, peripheral arterial disease, and/or cerebrovascular disease
* clinically relevant disease of the cardiovascular system, severe hepatic dysfunction (serum albumin <25 g/l or Child-Pugh score ≥10), severe renal dysfunction (estimated renal creatinine clearance <30 ml/min, clinical relevant disease of the nervous system, the endocrinium or another severe systematic disease
* Systemic lupus erythematodes or mixed connective tissue disease
* Inflammatory bowel disease
* alcohol or drug abuse during the last past 3 months
* Patients with hypertension BP persistently > 140/90mmHG) and has not been adequately controlled
* life expectancy <6 months
* state of mind which does not enable the patient to understand the nature of the study, its importance and possible consequences
* evidence that the respective person will not cooperate with the study protocoll
* participation of the patient in another clinical trial during the past 4 weeks before inclusion
* prior participation in this clinical trial

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss after implantation of a hip joint endoprosthesis | Three days
  The primary objective of the study is the designation of the perioperative blood loss after implantation of a hip joint endoprosthesis under the influence of Etoricoxib or of Diclofenac. The expectations hypothesis is that under Etoricoxib patients will loose a smaller quantity of blood than under Diclofenac.

SECONDARY OUTCOMES:
Heterotopic ossification | six months
  The secondary objectives are to investigate whether after hip joint endoprosthesis Etoricoxib can prevent heterotopic ossification in equal measure as Diclofenac
Postoperative pain | nine days
  It will be investigated if Diclofenac and Etoricoxib effectively reduce postoperative pain after hip joint endoprosthesis at rest and during movement.
Reduction of rescue medication | nine days
  It will be investigated whether Etioricoxib can reduce the use of rescue-medication as compared to Diclofenac
Gastroinstestinal tolerance | nine days
  It will be investigated if the gastrointestinal tolerance of Etoricoxib is superior to the one of Diclofenac

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic Surgery, Bad Abbach, Bavaria, Germany